CLINICAL TRIAL: NCT03286101
Title: A Randomized, Double-Blind, Placebo-Controlled Clinical Trial On The Efficacy And Safety Of Topical 0.5% Ivermectin Lotion For The Treatment Of Head Lice Infestation Among Filipino Children Age 3 Years Or Older
Brief Title: Efficacy and Safety of Topical 0.5% Ivermectin Lotion for the Treatment of Head Lice Infestation in Filipinos
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: United Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RD2017-01
Record Dates: First submitted 2017-09-14; First posted 2017-09-18 (Actual); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Pediculosis Capitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 0.5% Ivermectin Lotion (Experimental)
  Interventions: Drug: 0.5% Ivermectin lotion
- Vehicle control (Placebo Comparator)
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: 0.5% Ivermectin lotion — The intervention is composed of a single application of the 0.5% ivermectin lotion.
  Arms: 0.5% Ivermectin Lotion
Drug: Vehicle — The intervention is composed of a single application of the vehicle control.
  Arms: Vehicle control

SUMMARY:
This is a randomized, double-blind, placebo-controlled clinical study evaluating the efficacy and safety of a single application of 0.5% ivermectin lotion in Filipino subjects with head lice.

ELIGIBILITY:
Inclusion Criteria:

* Index subjects must have an active lice infestation defined as: At least 3 live lice (adult and/or nymphs) present on the scalp and/or hair as determined by a trained evaluator; After the index subject has been enrolled, additional infested household members will be enrolled.
* Household subjects must have an active head lice infestation defined as: At least 1 live louse (adult and /or nymph) present on the scalp and/or hair, as determined by a trained evaluator (with the exception of the male head of household who may self- assess, as being lice free).
* Subject is male or female;
* Subject is at least 3 years old or older at the time of enrollment;
* Subject is in good general health based on the medical history;
* Each adult subject must have an appropriately signed Informed Consent agreement. For children, parents/guardian must sign an Informed Parental Consent agreement for children not old enough to do so. Children of a specified age will be administered a child's assent form
* The caregiver of a subject must be willing to allow all household members to be screened for head lice. If other household members are found to have an active head lice infestation, they must be willing and able to participate in the study. No more than one working male per household maybe excluded from evaluation if he is assessed as being lice free by himself or the caregiver and cannot come in due to his work schedule. If this individual may have lice, he must come to the test facility, otherwise the entire household will be excluded from study participation.
* Subject and/or caregiver must be physically able and willing to report to the testing center for the supervised application of the product.
* Subjects agrees not to use any other form of lice treatment (commercial or mechanical/manual) while participating in the study;
* Following application and rinsing of the test product, subject agrees not to shampoo / wash, or rinse their hair or scalp until the 24-hour post treatment evaluation has been completed;
* Subject agrees to not cut or chemically treat their hair while participating in the study;
* Subject agrees to follow all study instructions.

Exclusion Criteria:

* History of irritation or sensitivity to ivermectin or lotion components pediculosis or hair care products;
* Presence of visible skin / scalp conditions that are not attributable to head lice infestation, such as erythema, blisters, vesicles which in the opinion of the investigative personnel will interfere with safety and / or efficacy evaluations;
* Subjects suffering from psoriasis, atopic dermatitis or other conditions, which in the opinion of the investigator may compromise the objective of the study;
* Treatment for head lice (OTC, home remedy or Rx) in the last 14 days;
* Subjects under treatment which in the opinion of the investigator will interfere with the study results;
* Subjects who participated in a previous investigational drug study within the past 30 days;
* Subjects who does not understand the requirements for the study participation and/ or likely exhibit poor compliance, in the opinion of the investigator;
* Females who are pregnant or lactating.
* Living in a household where at least one member is pregnant, lactating, or planning a pregnancy
* Subjects with skin lesions, specifically skin breaks are excluded because of possible absorption of the drug

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2017-09-14 (Actual); Primary Completion 2017-10-12 (Actual); Study Completion 2017-11-09 (Actual)

PRIMARY OUTCOMES:
Proportion of participants cured of head lice infestation from their assigned product on day 2, day 8 and day 15 after the first treatment. | Day 2 to day 15 after product application

CONTACTS AND LOCATIONS:
Overall Officials: Gertrude Chan, M.D., Principal Investigator — Clinical Trial Management and Testing Associates, Inc.
Locations (1):
- Clinical Trial Management and Testing Associates, Inc., City of Muntinlupa, Philippines

IPD SHARING:
Plan to Share IPD: No